CLINICAL TRIAL: NCT02528175
Title: Magnetic Resonance-Guided High Intensity Focused Ultrasound for Recurrent Rectal Cancer - A Pilot Study
Brief Title: Magnetic Resonance-Guided High Intensity Focused Ultrasound for Recurrent Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Chu, MD, MSc, FRCPC (Other)
Collaborators: Philips Medical Systems (Industry)
Responsible Party: Sponsor-Investigator, William Chu, MD, MSc, FRCPC, Radiation Oncologist, Clinician Investigator, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 273-2011; 226861 (Other: Health Canada)
Record Dates: First submitted 2015-06-09; First posted 2015-08-19 (Estimated); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Recurrent Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy; Drug Therapy; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRg-FU (Experimental): Hyperthermia via magnetic resonance-guided focused ultrasound will be administered once per week for three weeks concurrent with standard radiation and chemotherapy.
  Interventions: Device: Magnetic resonance-guided focused ultrasound; Radiation: Standard Radiation; Drug: Chemotherapy

INTERVENTIONS:
Device: Magnetic resonance-guided focused ultrasound — Targeted warming of the tumor via 3 weekly MR-guided ultrasound procedures. Concurrent with radiation and chemotherapy.
  Other Names: MRg-FU
Radiation: Standard Radiation — 30.6 Gray (Gy) over 17 fractions concurrent with chemotherapy (institutional standard).
  Other Names: Radiation Therapy
Drug: Chemotherapy — 3.5 weeks concurrent with radiation therapy (institutional standard).
  Other Names: Xeloda; Oral capecitabine

SUMMARY:
This pilot study hypothesizes that hyperthermia delivered via magnetic resonance-guided focused ultrasound (MRg-FU) is technically feasible and can be safely used in combination with concurrent reirradiation and chemotherapy for the treatment of recurrent rectal cancer. Twenty recurrent rectal cancer patients who are not candidates for surgery will be recruited for hyperthermia treatment delivered via MRg-FU concurrent with reirradiation and oral chemotherapy.

DETAILED DESCRIPTION:
Magnetic resonance-guided focused ultrasound (MRg-FU) is a non-invasive, outpatient modality being investigated for the thermal treatment of cancer. In MRg-FU, a specially designed transducer is used to focus a beam of low intensity ultrasound energy into a small volume at a specific target site in the body. MR is used to identify and delineate the tumour, focus the ultrasound beam on the target and provide real-time thermal mapping to ensure accurate heating of the designated target with minimal effect to the adjacent healthy tissue. The focused ultrasound beam produces therapeutic hyperthermia (40-42°C) in the target field causing protein denaturation and cell damage.

Currently, there is no prospective clinical data reported on the use of MRg-FU in the setting of recurrent rectal cancer. Recurrent rectal cancer is a vexing clinical problem. Current retreatment protocols have limited efficacy. The addition of hyperthermia to radiation and chemotherapy may enhance the therapeutic response. With recent advances in technology, the investigators hypothesize that MRg-FU is technically feasible and can be safely used in combination with concurrent reirradiation and chemotherapy for the treatment of recurrent rectal cancer without increased side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Weight <140kg
* Biopsy-proven recurrent rectal adenocarcinoma
* Assessed by the treating surgeon, medical oncologist and radiation oncologist, and following a multidisciplinary discussion, determined to have unresectable and/or inoperable disease in the presence or absence of distant metastases
* Assessed by the treating radiation oncologist and medical oncologist determined to be fit for reirradiation and chemotherapy
* Prior pelvic radiotherapy
* Target lesion visible by MR
* Target lesion accessible for MRg-FU procedure
* Target lesion maximum dimension ≤ 6cm
* Able to communicate sensation during MRg-FU treatment

Exclusion Criteria:

* Abdominal or pelvic surgery (excluding biopsy) ≤ 6 weeks prior to study enrolment
* Chemotherapy or other systemic anti-cancer agent ≤ 6 weeks prior to enrolment
* Previous radiotherapy ≤ 6 weeks prior to enrolment
* Recurrent tumour involves small bowel
* Unable to characterize pain
* Pregnant / Nursing woman
* Orthopaedic implant along proposed MRg-FU beam path or at site of target lesion.
* Serious cardiovascular, neurological, renal or hematological chronic disease
* Active infection
* Unable to tolerate required stationary position during treatment
* Allergy to MR contrast agent or sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-04; Primary Completion 2021-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Acute toxicities | 3 months
  Gastrointestinal and genitourinary toxicities assessed as per Common Toxicity Criteria for Adverse Effects (CTCAE) v4.0 after each MRg-FU treatment and 30, 60 and 90 days post-treatment.

SECONDARY OUTCOMES:
Late toxicities | 3 years
  Gastrointestinal and genitourinary toxicities assessed as per CTCAE v4.0 every 6 months post-treatment for three years.
The efficacy of MRg-FU in reducing pain | 3 years
  Patient reported pain will be assessed through completion of the Brief Pain Inventory (BPI) and reporting of analgesic usage after each MRg-FU treatment, monthly post-treatment for three months and every 6 months post-treatment for 3 years.
Patient quality of life | 3 years
  Patient reported quality of life will be assessed through completion of the European Organization for Research and Treatment of Cancer (EORTC) Functional Assessment of Cancer Therapy - Colorectal (FACT-C) questionnaire after each MRg-FU treatment, monthly post-treatment for three months and every 6 months post treatment for 3 years.
Assessment of radiologic response following treatment. | 3 years
  Assessment of response using the EORTC Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: William Chu, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Peng J, Partanen A, Pichardo S, Staruch R, Perry K, McGuffin M, Huang Y, Chan KK, Wong S, Czarnota G, Hynynen K, Chu W. Mild hyperthermia with magnetic resonance- guided high intensity focused ultrasound combined with salvage chemoradiation for recurrent rectal cancer. Int J Hyperthermia. 2024;41(1):2365385. doi: 10.1080/02656736.2024.2365385. Epub 2024 Jun 19. PMID 38897584